CLINICAL TRIAL: NCT00902421
Title: Efficacy and Safety of SSRI in Overactive Bladder Patients; a 3-month, Prospective, Open-label, Comparative Study
Brief Title: Efficacy and Safety of Selective Serotonin Reuptake Inhibitor (SSRI) in Overactive Bladder Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Kyu-Sung Lee/Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-08-047
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2010-08-26 (Estimated); Status verified 2010-08

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; SSRI; Antimuscarinics
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Selective Serotonin Reuptake Inhibitors; Escitalopram; Muscarinic Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antimuscarinics (Active Comparator)
  Interventions: Drug: Antimuscarinics
- Selective serotonin reuptake inhibitors (Experimental): Selective serotonin reuptake inhibitor
  Interventions: Drug: Selective serotonin reuptake inhibitors

INTERVENTIONS:
Drug: Selective serotonin reuptake inhibitors — escitalopram 10mg once daily for 3 months
  Other Names: Lexapro®
  Arms: Selective serotonin reuptake inhibitors
Drug: Antimuscarinics — Antimuscarinics for 3 months
  Arms: Antimuscarinics

SUMMARY:
The urologic literature suggests that there is an association between a variety of psychiatric disorders and incontinence. Most notably, depression is found in a significant percentage of patients with urinary incontinence. Depression also occurs in other conditions associated with urinary urge incontinence, such as aging and dementia, and in neurologic disorders such as normal pressure hydrocephalus. Correction of some neurologic disorders eliminates both depression and urge incontinence. Although chronic medical disorders such as urge incontinence may lead to depression, an alternative hypothesis is that these two conditions share a common neurochemical pathogenesis. Lowering monoamines such as serotonin and noradrenaline in the central nervous system (CNS) leads to depression and urinary frequency and a hyperactive bladder in experimental animals. Thus, depression may not only be the result of persistent urinary incontinence, but individuals with altered CNS monoamines could manifest both depression and an overactive bladder. The latter condition may lead to urge incontinence, urinary frequency, urgency, or enuresis. Uncovering further evidence for such a linkage could serve as the basis for the development of genetic markers and novel therapeutic interventions for these two conditions.

In this study, the investigators will evaluate the efficacy and safety of SSRI on OAB patients who does not respond to the antimuscarinic agents.

DETAILED DESCRIPTION:
* 3-month, prospective, open-label, comparative trial
* Primary Objectives:

  * To investigate the changes of OAB symptoms in patients who did not showed therapeutic benefits after 3 months of treatment with antimuscarinic agents and who then treated with SSRI (escitalopram) for 3 months.
* Secondary Objectives

  * To investigate the change of patient perception of urgency and bladder condition
  * To investigate the change of patient perception of quality of life
  * To investigate the change of psychologic parameters
  * To investigate the patient perception of treatment benefit
  * To find the predictive factors of patients who respond to the 3 month-treatment with escitalopram
  * To explore the efficacy of escitalopram on the tolerability and safety

ELIGIBILITY:
Inclusion Criteria:

* Female aged ≥ 18 and ≤80 years
* On a stable dose of an antimuscarinic agents for at least 3 months
* Persistent symptoms of OAB as verified by the screening 5 day micturition diary, defined by:

  1. Mean urinary frequency ≥8 times/24 hours
  2. Mean number of urgency episodes, with/without urgency incontinence, ≥1 episode/24 hours (with a Urinary Sensation Scale rating of ≥3 in the micturition diary)
* A rating of the bladder condition at Baseline prior to randomization as "Some Moderate Problems", "Severe Problems", or "Many Severe Problems" on the Patient Perception of Bladder Condition (PPBC) questionnaire
* Ability and willingness to correctly complete the micturition diary and questionnaire
* Capable of understanding and having signed the informed consent form after full discussion of the research nature of the treatment and its risks and benefits

Exclusion Criteria:

* Clinical significant stress incontinence as determined by the investigator and confirmed for female patients by a cough provocation test
* An average volume voided of > 200 ml per micturition as verified on the baseline micturition diary
* Total daily urine volume of > 3000 ml as verified on the baseline micturition diary
* Patients who have past psychiatric disease such as major depression, anxiety disorder, panic disorder, and so on.
* Significant hepatic or renal disease, defined as having twice the upper limit of the reference ranges for serum concentrations of aspartate aminotransferase (AST [SGOT]), alanine aminotransferase (ALT [SGPT]), alkaline phosphatase or creatinine
* Any condition that is a contraindication for anticholinergic treatment, including uncontrolled narrow-angled glaucoma, urinary retention or gastric retention
* Symptomatic acute urinary tract infection (UTI) during the run-in period
* Recurrent UTIs defined as having been treated for symptomatic UTIs > 4 times in the last year
* Diagnosed or suspected interstitial cystitis
* Uninvestigated hematuria or hematuria secondary to malignant disease
* Clinically significant bladder outlet obstruction defined by clinical symptoms and investigator's opinion according to local standard of care
* Patients with marked cystocele or other clinically significant pelvic prolapse.
* On an unstable dosage of any drug with anticholinergic side effects, or expected to start such treatment during the study
* Receipt of any electrostimulation or bladder training within the 14 days before the start of tolterodine SR, or expected to start such treatment during the study
* An indwelling catheter or practicing intermittent self-catheterization Use of any investigational drug within 2 months preceding the start of the study
* Patients with chronic constipation or history of severe constipation
* Pregnant or nursing women
* Sexually active females of childbearing potential not using reliable contraception for at least 1 month prior to study start and not agreeing to use such methods during the entire study period and for at least 1 month thereafter. Reliable contraceptive methods are defined as intrauterine devices (IUDs), combination type contraceptive pills, hormonal implants, double barrier method, injectable contraceptives and surgical procedures (tubal ligation or vasectomy).
* Patients who have bladder cancer
* Use of any nonselective, irreversible MAO inhibitor
* Any other condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Percentage change in urgency episodes/24 hrs | 3 months of medication

SECONDARY OUTCOMES:
Micturition diary efficacy parameters | 3 months of medication
Quality of life parameters | 3 months of medication
Patient perceptions | 3 months of medication
Psychologic parameters | 3 months of medication

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea